CLINICAL TRIAL: NCT02250014
Title: The Immuno-Response to Primary Cryotherapy for the Treatment of Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0071.cc; 14-0071 (Other: University of Colorado, Denver)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryotherapy; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cryotherapy, sargramostim) (Experimental): Patients undergo cryotherapy on day 0 and receive sargramostim subcutaneously on days 1, 3, 5, 8, 10, and 12.
  Interventions: Procedure: cryotherapy; Biological: sargramostim
- Arm II (cryotherapy, standard of care) (Active Comparator): Patients undergo cryotherapy on day 0.
  Interventions: Procedure: cryotherapy

INTERVENTIONS:
Procedure: cryotherapy — Undergo cryotherapy
Biological: sargramostim — Given subcutaneously
  Other Names: GM-CSF; Leukine; Prokine
  Arms: Arm I (cryotherapy, sargramostim)

SUMMARY:
This randomized pilot phase I trial studies how well sargramostim after cryotherapy works in treating patients with prostate cancer. Biological therapies, such as sargramostim, use substances made from living organisms that may stimulate the immune system in different ways and stop tumor cells from growing. Cryosurgery, also known as cryotherapy, kills tumor cells by freezing them. Giving sargramostim after cryotherapy may work better in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine an unknown normal immune response (T cell and B cell) to post-cryotherapy treatment for prostate cancer.

II. Detect the altered immune response (T cell and B cell) post-GM-CSF (sargramostim) response and post-cryotherapy for the prostate cancer.

Patients are randomized to 1 of 2 treatment arms.

ARM I (TREATMENT): Patients undergo cryotherapy on day 0 and receive sargramostim subcutaneously (SC) on days 1, 3, 5, 8, 10, and 12.

ARM II (CONTROL): Patients undergo cryotherapy on day 0.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with prostate cancer that elect to undergo primary cryotherapy of the prostate
* Patients who are diagnosed with clinical stage T1a -T2c prostate cancer
* Gleason score sum of less than or equal to 7
* Prostate-specific antigen (PSA) < 20 ng/dl
* Patient will read, understand and sign the informed consent and Health Insurance Portability and Accountability Act (HIPAA) agreement
* Patients must have a life expectancy of at least one year

Exclusion Criteria:

* Known hypersensitivity to granulocyte macrophage colony stimulating factor (GM-CSF) or yeast
* Anticipated blood donation within the next 90 days
* Magnetic resonance imaging (MRI), computed tomography (CT) and bone scan evidence of metastatic prostate cancer regardless the PSA level; (the indication for which is clinically driven and at the discretion of the treating physician)
* Any history of current or within the past 48 hours of acute or chronic bacterial, fungal or viral infectious disease
* Documented excessive leukemic myeloid blasts in the bone marrow or peripheral blood (>= 10%) in the past 6 months
* Previous organ transplant
* Immunosuppression including primary, secondary, iatrogenic and idiopathic
* Other serious diseases (hematological, hepatic, renal, respiratory, central nervous system, autoimmune or psychiatric)
* Enrollment in other studies for any disease in the past 30 days
* Diagnosis of cancer that in not considered cured, except basal cell carcinoma (BCC) of skin
* Prior transurethral resection of the prostate with a large tissue defect (at the discretion of the investigator)
* History of abdominoperineal resection for rectal cancer, rectal stenosis, or other major rectal pathology
* Patient currently receiving lithium, steroid, chemotherapy or radiotherapy treatment
* Patients with a Hemoglobin of less than 12%

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Change in B cell response identified by Serametrix assay | Baseline to up to 3 months after cryotherapy
  A scatter plot of each cytokine and antigen level will be created for each patient by marker to observe the behavior of the markers (rising, falling, flat, or combination over time). Patient specific pre-operative levels will be used to obtain individual baseline measures from which the difference in follow-up cytokine and antigen levels will be calculated, then a simple descriptive comparison of the mean elevation in the markers' levels across cohorts will be graphed.
Change in T cell responses identified by Intracellular cytokine assay and enzyme-linked immunospot | Baseline to up to 3 months after cryotherapy
  A scatter plot of each cytokine and antigen level will be created for each patient by marker to observe the behavior of the markers (rising, falling, flat, or combination over time). Patient specific pre-operative levels will be used to obtain individual baseline measures from which the difference in follow-up cytokine and antigen levels will be calculated, then a simple descriptive comparison of the mean elevation in the markers' levels across cohorts will be graphed.

SECONDARY OUTCOMES:
Change in PSA levels in serum samples | Up to 6 months after cryotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Al Barqawi, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No